CLINICAL TRIAL: NCT02144181
Title: Evaluation of the Safety and Efficacy of the Ulthera® System for the Treatment of Signs and Symptoms of Erythematotelangiectatic Rosacea
Brief Title: Ultherapy® for the Treatment of Erythematotelangiectatic Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-138
Record Dates: First submitted 2014-05-19; First posted 2014-05-21 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2016-10

CONDITIONS: Erythematotelangiectatic Rosacea; Rosacea
Keywords: Ulthera® System; Ultherapy® Treatment; Ulthera, Inc.
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A (Active Comparator): Subjects will receive two low-density Ulthera System Treatments. Protocol amended Sept 2014: Subjects will receive one low-density Ulthera System Treatment.
  Interventions: Device: Ulthera System Treatment
- Group B (Active Comparator): Subjects will receive three low-density Ulthera System Treatments. Protocol amended Sept 2014: Subjects will receive two low-density Ulthera System Treatments.
  Interventions: Device: Ulthera System Treatment
- Group C (Active Comparator): Subjects will receive two high-density Ulthera System Treatments. Protocol amended Sept 2014: Subjects will receive one high-density Ulthera System Treatment.
  Interventions: Device: Ulthera System Treatment
- Group D (Active Comparator): Subjects will receive three high-density Ulthera System Treatments. Protocol amended Sept 2014: Subjects will receive two high-density Ulthera System Treatments.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy®

SUMMARY:
This is a prospective, multi-site (up to 5 sites), single-blinded, randomized trial. Up to 88 subjects will be enrolled and randomized to one of four treatment groups (4 Groups of 22 subjects), and will receive study treatments based on their assigned treatment group. Following study treatments, follow-up visits will occur at 90, 180 and 365 days from each subject's last study treatment.

DETAILED DESCRIPTION:
Clinician Erythema Assessment (CEA) and Patient Self-Assessment (PSA) scores, assessing severity of erythema, will be obtained prior to study treatment to confirm subject eligibility. Enrolled subjects will receive up to three dual-depth treatments to affected areas of the midface (cheeks, chin, forehead, glabella and nose) each treatment provided approximately 2 weeks apart. Groups A and B will receive low-density treatment, and Groups C and D receive high-density treatment. Groups A and C will receive 2 treatments. Groups B and D will receive 3 treatments. Protocol amended Sept 2014: Groups A and C will receive 1 treatment; Groups B and D will receive 2 treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 65 years.
2. Subject in good health.
3. Clinical diagnosis of Erythematotelangiectatic Rosacea.
4. Understands and accepts the obligation not to undergo any other elective procedures, i.e., laser and IPL, in the areas to be treated through the follow-up period.
5. A Clinician Erythema Assessment (CEA) score of greater than or equal to 3 at Screening and at Baseline/Day 0 (prior to study treatment commencement).
6. A Patient Self-Assessment (PSA) of erythema score of greater than or equal to 2 at Screening and at Baseline/Day 0 (prior to study treatment commencement).
7. Willingness to refrain from use of aspirin, Ibuprofen, Naproxen or any other NSAID prior to each study treatment and chronic use during the entire post-treatment study period. Washout period, if chronic user, for 4 weeks prior to the first treatment. After all study treatments are completed, limited acute NSAID use is allowed. A maximum of 2-3 doses, in the 2 weeks prior to study follow-up visits is allowed, if needed.
8. Willingness to continue using current skin care and topical treatment regimen during the entire study period (1 year).
9. Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study, unless deemed medically necessary.
10. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control .
11. Absence of physical or psychological conditions unacceptable to the investigator.
12. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
13. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active systemic disease that may affect wound healing.
2. More than 5 prominent telangiectases (>0.2mm in width, the width of a thick human hair, images will be provided) in the area(s) to be treated, with the exception of the lateral sides of the nose.
3. Particular forms of rosacea (papulopustular, phymatous, ocular Rosacea, rosacea conglobata, rosacea fulminans, isolated rhinophyma, isolated pustulosis of the chin) or other concomitant facial dermatoses that are similar to rosacea such as peri-oral dermatitis, demodicidosis, facial keratosis pilaris, seborrheic dermatitis, or acute lupus erythematosus.
4. Presence of three (3) or more facial inflammatory lesions (papules or pustules) of rosacea.
5. Current treatment with monoamine oxidase (MAO) inhibitors, barbiturates, opiates, sedatives, systemic anesthetics, or alpha agonists.
6. Intense flushing to a few triggers, such as post-menopausal hot flashes or particular food, versus both intense and less intense flushing to several common triggers.
7. Less than 3 months stable dose treatment with tricyclic anti-depressants, cardiac glycosides, beta blockers or other antihypertensive agents which have vasodilation as the MOA (e.g., the calcium channel blockers, such as nifedipine).
8. Current diagnosis of Raynaud's syndrome, thromboangiitis obliterans, orthostatic hypotension, severe cardiovascular disease, cerebral or coronary insufficiency, renal or hepatic impairment, scleroderma, Sjögren's syndrome, or clinically diagnosed depression (unless on a stable treatment regimen.)
9. History of post-inflammatory hyperpigmentation.
10. Severe solar elastosis.
11. Significant scarring that would interfere with assessing results in areas to be treated.
12. Open wounds or lesions in the area(s) to be treated.
13. Acne.
14. Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included.)
15. Inability to understand the protocol or to give informed consent.
16. Microdermabrasion or glycolic acid peels to the treatment areas within four weeks prior to study participation or during the study.
17. Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
18. History of chronic drug or alcohol abuse.
19. History of autoimmune disease.
20. History of Bell's Palsy or epilepsy
21. History of diabetes.
22. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
23. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
24. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
25. Concurrent enrollment, or participated within the past 30 days, in any study involving the use of investigational devices or drugs.
26. Current smoker or history of smoking in the last five years.
27. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
28. History of the following cosmetic treatments in the areas to be treated:

    1. Skin tightening procedure within the past year;
    2. Injectable filler of any type within the past:

    i. 12 months for Hyaluronic acid fillers (e.g.,Restylane)

    ii. 12 months for Ca Hydroxyapatite fillers (e.g., Radiesse)

    iii. 24 months for Long-lasting Hyaluronic acid (Juvéderm Voluma) and Poly-L-Lactic acid fillers (e.g., Sculptra)

    iv. Ever for permanent fillers (e.g., Silicone, ArteFill)

    c. Neurotoxins within the past three months;

    d. Ablative resurfacing laser treatment;

    e. Nonablative, rejuvenative laser or light treatment within the past six months;

    f. Surgical dermabrasion or deep facial peels;
29. History of using Accutane or other systemic retinoids within the past six months;
30. Topical retinoids within the past two weeks;
31. Antiplatelet agents / Anticoagulants (Coumadin, Heparin, Plavix);
32. Chronic use of non-steroidal anti-inflammatories (naproxen, ibuprofen, etc.) within the past 4 weeks.
33. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements, understanding and signing the informed consent, or affect their ability to accurately complete QOL and subjective improvement assessments.
34. Use of Mirvaso (topical brimonidine tartrate) within the previous two weeks.
35. Use of systemic corticosteroid or immunosuppressive drugs.
36. Use of antipruritics, including antihistamines, within 24 hours of study visits.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Clinician Erythema Assessment at 90 days post-treatment compared to baseline | 90 Days post-treatment
  Erythema will be assessed on a 5-point Clinician Erythema Assessment (CEA) scale (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) at baseline and at 90 days post-treatment completion. Success is defined as 1-grade improvement on CEA scale.

SECONDARY OUTCOMES:
CEA scale at 180 days post-treatment compared to baseline. | 180 Days post-treatment
  Erythema will be assessed on a 5-point Clinician Erythema Assessment (CEA) scale (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) at baseline and at 180 days post-treatment completion.
CEA scale at 365 days post-treatment compared to baseline. | 365 Days post-treatment
  Erythema will be assessed on a 5-point Clinician Erythema Assessment (CEA) scale (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) at baseline and at 365 days post-treatment completion.
Patient Self-Assessment (PSA) of erythema at 90 Days compared to baseline. | 90 Days post-treatment
  Patient Self-Assessment (PSA) of erythema (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) completed at 90 Days post-treatment.
Patient Self-Assessment (PSA) of erythema at 180 Days compared to baseline. | 180 Days post-treatment
  Patient Self-Assessment (PSA) of erythema (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) completed at 180 Days post-treatment.
Patient Self-Assessment (PSA) of erythema at 365 Days compared to baseline. | 365 Days post-treatment
  Patient Self-Assessment (PSA) of erythema (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe) completed at 365 Days post-treatment.
Dermatology Life Quality Index (DLQI) Assessment at 90 Days post-treatment | 90 Days post-treatment
  Dermatology Life Quality Index (DLQI) Assessment at 90 Days post-treatment compared to baseline, a 10-question validated questionnaire.
Dermatology Life Quality Index (DLQI) Assessment at 180 Days post-treatment | 180 Days post-treatment
  Dermatology Life Quality Index (DLQI) Assessment at 180 Days post-treatment compared to baseline, a 10-question validated questionnaire.
Dermatology Life Quality Index (DLQI) Assessment at 365 Days post-treatment | 365 Days post-treatment
  Dermatology Life Quality Index (DLQI) Assessment at 365 Days post-treatment compared to baseline, a 10-question validated questionnaire.
Colorimeter at 90 Days post-treatment | 90 Days post-treatment
  Colorimeter at 90 Days post-treatment compared to baseline. An objective evaluation of the intensity of erythema as a measure of redness using a colorimeter.
Colorimeter at 180 Days post-treatment | 180 Days post-treatment
  Colorimeter at 180 Days post-treatment compared to baseline. An objective evaluation of the intensity of erythema as a measure of redness using a colorimeter.
Colorimeter at 365 Days post-treatment | 365 Days post-treatment
  Colorimeter at 365 Days post-treatment compared to baseline. An objective evaluation of the intensity of erythema as a measure of redness using a colorimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lupin, MD, Principal Investigator — Cosmedica Laser Centre
Locations (5):
- United States (4):
  - Skin Specialists, PC, Omaha, Nebraska
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - All About Faces, Hummelstown, Pennsylvania
  - Laser & Cosmetic Center, Virginia Beach, Virginia
- Cosmedica Laser Centre, Victoria, British Columbia, Canada